CLINICAL TRIAL: NCT00371709
Title: TAXUS ATLAS: A Multi-center, Single-arm Study of the TAXUS Liberté™-SR Stent for the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: TAXUS ATLAS: TAXUS Liberté™-SR Stent for the Treatment of de Novo Coronary Artery Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2013; TAXUS ATLAS
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Liberté-SR
- Arm 2 (Other): Historical Comparator: control data derived from the TAXUS IV and TAXUS V studies
  Interventions: Device: TAXUS™ Express

INTERVENTIONS:
Device: TAXUS Liberté-SR — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 1
Device: TAXUS™ Express — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 2

SUMMARY:
TAXUS ATLAS is a global, multi-center, single-arm, non-inferiority trial comparing results from patients treated with the TAXUS Liberté stent to an historical TAXUS Express control. The control group is a case-matched, blended population of TAXUS Express patients from the TAXUS IV and TAXUS V de novo clinical trials. The objective of the study is to evaluate clinical outcomes of TAXUS Liberté-SR stent in de novo lesions and to assess the non-inferiority of TAXUS Liberté versus TAXUS Express. The TAXUS Liberté-SR stent is hypothesized to have comparable safety and efficacy to the TAXUS Express stent.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient is ≥18 years old.
2. Eligible for percutaneous coronary intervention (PCI)
3. Documented stable angina pectoris or unstable angina pectoris with documented ischemia or documented silent ischemia
4. Left ventricular ejection fraction (LVEF) of >/=25%
5. Acceptable candidate for coronary artery bypass grafting (CABG)
6. Patient or legal guardian understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
7. Willing to comply with all specified follow-up evaluations

Angiographic Inclusion Criteria:

1. Only one lesion (target lesion) may be treated with the study stent. However, one additional lesion in a non-target vessel may be treated during the index procedure with a commercially available bare metal stent, heparin-coated stent or TAXUS Express stent.
2. Target lesion enrolled for treatment may be composed of multiple lesions (not more than 10mm between diseased segments)but must be completely covered by one study stent.
3. Target lesion located within a single native coronary artery
4. Cumulative target lesion length is ≥10 mm and ≤28 mm (visual estimate)
5. RVD of ≥2.5 mm to ≤4.0 mm (visual estimate)
6. Target lesion diameter stenosis ≥50% (visual estimate)
7. Target lesion is de novo (i.e., a coronary lesion not previously treated)

General Exclusion Criteria:

1. Known hypersensitivity to paclitaxel
2. Any previous, concurrent or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent.
3. Previous or planned use of both the study stent and a non-study stent (i.e., commercial stent) in the treatment of the target vessel
4. Previous or planned treatment with intravascular brachytherapy in the target vessel
5. Planned CABG ≤9-months post-index procedure
6. MI within 72 hours prior to the index procedure and or creatine kinase(CK) >2x the local laboratory's ULN unless CK-MB is <2x ULN.
7. Cerebrovascular Accident (CVA) within the past 6 months
8. Cardiogenic Shock
9. Acute or chronic renal dysfunction
10. Contraindication to ASA, or to both clopidogrel and ticlopidine
11. Leukopenia
12. Thrombocytopenia or thrombocytosis
13. Active peptic ulcer or active gastrointestinal (GI) bleeding
14. Known allergy to stainless steel
15. Any prior true anaphylactic reaction to contrast agents
16. Patient is currently, or has been treated with paclitaxel or other chemotherapeutic agents within 12-months of the index procedure
17. Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9-months after the index procedure
18. Male or female with known intention to procreate within 3 months after the index procedure
19. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the study.
20. Life expectancy of less than 24-months due to other medical condition
21. Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
22. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Angiographic Exclusion Criteria:

1. Left main coronary artery disease (stenosis >50%) whether protected or unprotected
2. Target lesion is ostial in location (within 3.0 mm of vessel origin)
3. Target lesion and/or target vessel proximal to the target lesion is moderately or severely calcified by visual estimate.
4. Target lesion and/or target vessel proximal to the target lesion is tortuous.
5. Target lesion is located within or distal to a >60 degree bend in the vessel
6. Target lesion involves a bifurcation with a side branch vessel >2.0 mm in diameter.
7. Target lesion is totally occluded (TIMI flow </= 1), either at baseline or predilation
8. Angiographic presence of probable or definite thrombus
9. Pre-treatment of the target vessel is not allowed with any device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 871 (Actual)
Dates: Start 2004-08; Primary Completion 2005-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
9-Month Target Vessel Revascularization (TVR) | 9 Months

SECONDARY OUTCOMES:
Clinical procedural and technical success | 5 Years
Utilization parameters (equipment utilization; catheters, guidewires and balloons, procedure time, fluoroscopic time and amount of contrast used) | 9 Months
MACE rates at discharge, 1, 4 and 9-months and 1, 2, 3, 4, and 5 years post-index procedure. | 5 Years
Stent thrombosis rate | 5 Years
Target Vessel Failure (TVF) | 5 Years
QCA parameters (binary restenosis rate, MLD and late loss) | 9 Months
IVUS parameters (percent net volume obstruction, incomplete apposition, stent and area volumes, neointimal area volume) for patients in the IVUS subset | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Turco, MD, Principal Investigator — Washington Adventist Hospital; John A Ormiston, MD, Principal Investigator — Mercy Hospital; Peter Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (62):
- United States (40):
  - Baptist Medical Center Princeton Cardiology PC, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Brotman Medical Center, Beverly Hills, California
  - Mercy General Hospital, Sacramento, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - University of California San Diego Medical Center, San Diego, California
  - St. Joseph's Medical Center, Stockton, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Christiana Hospital, Newark, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Rockford Cardiology Associates, Rockford, Illinois
  - Praire Cardiovascular Consultants, Ltd., Springfield, Illinois
  - The Heart Center, Indianapolis, Indiana
  - Willis Knighton Medical Center, Shreveport, Louisiana
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Dartmouth Hitchcock Cardiology, Lebanon, New Hampshire
  - New York Presbyterian Hospital, New York, New York
  - WakeMed, Raleigh, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - North Ohio Research Elyria Memorial Hospital, Elyria, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - The Pennsylvania State University Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Methodist DeBakey Heart Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - St. Peter Hospital, Olympia, Washington
  - Northwest Cardiovascular Research Institute-Spokane Cardiology, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Aurora St Lukes Medcial Center, Milwaukee, Wisconsin
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Cardiovascular Research Center Monash Medical Centre, Clayton, Victoria
  - Epworth Hospital, Richmond, Victoria
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM Notre-Dame Hospital, Montreal, Quebec
- Queen Elizabeth Hospital, Kowloon, China
- New Zealand (4):
  - Mercy Angiography Unit, 98 Mountain Road, First Floor, Auckland, Epsom
  - Christchurch Hospital, Christchurch, New Zealand
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
- Taiwan (6):
  - Chang-Gung Memorial Hospital, Kaohsiung, Dawan
  - Shin Kong Memorial Hospital, Shih Lin Taipei 111
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Linkou, Taoyuan District

REFERENCES:
- [Derived] Ormiston JA, Charles O, Mann T, Hall JJ, McGarry T, Cannon LA, Webster MW, Mishkel GJ, Underwood PL, Dawkins KD. Final 5-year results of the TAXUS ATLAS, TAXUS ATLAS Small Vessel, and TAXUS ATLAS Long Lesion clinical trials of the TAXUS Liberte paclitaxel-eluting stent in de-novo coronary artery lesions. Coron Artery Dis. 2013 Jan;24(1):61-8. doi: 10.1097/MCA.0b013e32835b3932. PMID 23232250
- [Derived] Mahmud E, Ormiston JA, Turco MA, Popma JJ, Weissman NJ, O'Shaughnessy CD, Mann T, Hall JJ, McGarry TF, Cannon LA, Webster MW, Mandinov L, Baim DS. TAXUS Liberte attenuates the risk of restenosis in patients with medically treated diabetes mellitus: results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2009 Mar;2(3):240-52. doi: 10.1016/j.jcin.2008.12.009. PMID 19463432
- [Derived] Turco MA, Ormiston JA, Popma JJ, Mandinov L, O'Shaughnessy CD, Mann T, McGarry TF, Wu CJ, Chan C, Webster MW, Hall JJ, Mishkel GJ, Cannon LA, Baim DS, Koglin J. Polymer-based, paclitaxel-eluting TAXUS Liberte stent in de novo lesions: the pivotal TAXUS ATLAS trial. J Am Coll Cardiol. 2007 Apr 24;49(16):1676-83. doi: 10.1016/j.jacc.2007.01.069. Epub 2007 Apr 6. PMID 17448368